CLINICAL TRIAL: NCT03776006
Title: Registry of Transperineal Laser Ablation for Treatment of Lower Urinary Tract Symptoms With Use of the Echolaser® Device: A Multicentre, International Registry to Evaluate the Treatment of LUTS in Terms of Long-term Efficacy, Functional Outcomes and Safety
Brief Title: Registry: TPLA for LUTS
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. T.M. de Reijke, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W18_316
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostate Hyperplasia; Benign Prostatic Hypertrophy With Outflow Obstruction
Keywords: Transperineal laser ablation; LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TPLA
  Interventions: Procedure: Transperineal Laser Ablation

INTERVENTIONS:
Procedure: Transperineal Laser Ablation — Transperineal Laser Ablation of the Prostate
  Other Names: Echolaser X4

SUMMARY:
Rationale: The treatment of lower urinary tract symptoms (LUTS) due to benign prostatic enlargement in men with transperineal laser ablation (TPLA) may offer advantages in functional outcomes and safety over current standard therapies. As the technique is relatively new, indications and outcomes for this treatment are subject of investigation. However, the technique is already applied outside clinical studies. Clinical information from these treatments can be useful for future research. The aim of this study is to collect data on patients treated with transperineal laser ablation of the prostate outside clinical trials and to provide data on safety and functional outcomes in these patients in order to improve treatment.

Objective: To assess long-term efficacy of transperineal laser ablation for lower urinary tract symptoms, to assess functional outcomes, to assess safety, to determine baseline patient characteristics, to collect information on possible differences between centres applying treatment of transperineal laser ablation and to explore the optimal treatment indications and possible limitations.

Study design: This is an international prospective observational study in which data is recorded of patients who are treated with transperineal laser ablation for lower urinary tract symptoms.

Study population: Male patients treated with transperineal laser ablation for lower urinary tract symptoms due to benign prostatic enlargement.

Main study parameters/endpoints: The primary endpoint of this study is long-term efficacy of transperineal laser ablation for lower urinary tract symptoms measured by the time until surgical retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Presenting with lower urinary tract symptoms
* Indication for transperineal laser ablation
* Signed informed consent form

Exclusion Criteria:

* Age < 18 years
* Previous or active treatment for prostate cancer (active surveillance is not seen as active treatment)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises those patients presenting with lower urinary tract symptoms due to benign prostatic enlargement and are planned to undergo transperineal laser ablation in the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Long-term treatment efficacy measured by the time until surgical retreatment. | 5 years following TPLA treatment
  The treatment effectiveness is measured by the time until the need for surgical retreatment. This is measured by the time between the TPLA treatment and retreatment indicated due to new micturion problems. The time is expressed in years.

SECONDARY OUTCOMES:
Experienced functional efficacy measured by change in International Prostate Symptom Score | 12 months following TPLA treatment
  The experienced functional efficacy is measured by change in the International Prostate Symptom Score (IPSS). The IPSS is a is a self-administered scale of 7 questions concerning urinary symptoms plus one question concerning quality of life (QoL). Each of the seven symptoms includes the assignment of scores from 0 to 5. The total score can therefore range from 0 to 35 points (asymptomatic to very symptomatic). The patient's quality of life (QoL) will be evaluated separately.
Objectified functional efficacy measured by change of maximum flow by uroflowmetry. | 12 months following TPLA treatment
  Change in maximum urinary flow rate after 12 months compared to baseline.
Long-term treatment efficacy measured by the time until restart of urological medication. | 5 years following TPLA treatment
  The treatment effectiveness is measured by the time until the need for medical treatment due to new miction symptoms. This is measured by the time between the TPLA treatment and start of medical treatment for LUTS. The time is expressed in years.
Procedural safety measuered by the incidence of TPLA procedure related adverse events, reported by the CTCAE v5.0.. | 1 day following TPLA treatment
  Number of intraoperative adverse events using the CTCAE v5.0. Procedural safety is shown when no adverse events of grade 3 or higher.
Treatment safety measured by adverse event incidence at 30 days, reported by the CTCAE v5.0 | 30 days following TPLA treatment
  Number of adverse events using the CTCAE v5.0. Treatment safety is shown when no adverse events of grade 3b or higher are reported at 30 days post-TPLA treatment.

IPD SHARING:
Plan to Share IPD: Undecided